CLINICAL TRIAL: NCT05994391
Title: A Prospective, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Effects of LasoperinTM on Cognitive Function in Healthy Adults
Acronym: COG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lindenwood University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IRB-22-78
Record Dates: First submitted 2023-08-08; First posted 2023-08-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Cognitive Impairment; Cognitive Decline; Cognition Disorders in Old Age; Well-Being, Psychological; Inflammation; Cognitive Fun
Keywords: cognitive function; inflammation; well being
MeSH Terms: conditions — Cognitive Dysfunction; Psychological Well-Being; Inflammation

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, parallel design
Who Masked: Participant, Investigator
Masking Description: All supplements will be in sealed, blinded packaging with identical information on each package. Supplements will be blinded by a third party who is not a member of the research team.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LasoperinTM (Experimental): Active ingredients:
  Scutellaria baicalensis extract, 240 mg per capsule. Acacia catechu extract, 51 mg per capsule. With no less than 180 mg of baicalin, and no less than 30 mg of catechins from the above-mentioned extracts per capsule.
  Inactive ingredients:
  Maltodextrin
  2 capsules per day
  Take twice per day with food and water, once in the morning and once in the evening.
  If a dose is missed the participant can consume it as soon as they remember within the day. This means that the participant may consume 2 capsules at once. If both capsules are missed for the day the participant should not consume 4 capsules the next day and should return to the normal dosage of one capsule in the morning and evening
  Interventions: Dietary Supplement: LasoperinTM
- Placebo (Placebo Comparator): Active ingredients:
  N/A
  Inactive ingredients:
  Microcrystalline cellulose
  2 capsules per day
  Take twice per day with food and water, once in the morning and once in the evening.
  If a dose is missed the participant can consume it as soon as they remember within the day. This means that the participant may consume 2 capsules at once. If both capsules are missed for the day the participant should not consume 4 capsules the next day and should return to the normal dosage of one capsule in the morning and evening
  Interventions: Dietary Supplement: Placeo

INTERVENTIONS:
Dietary Supplement: LasoperinTM — Active ingredients:
  Scutellaria baicalensis extract, 240 mg per capsule. Acacia catechu extract, 51 mg per capsule. With no less than 180 mg of baicalin, and no less than 30 mg of catechins from the above-mentioned extracts per capsule.
  Inactive ingredients:
  Maltodextrin
  Arms: LasoperinTM
Dietary Supplement: Placeo — Active ingredients:
  N/A
  Inactive ingredients:
  Microcrystalline cellulose
  Arms: Placebo

SUMMARY:
The potential impact of various dietary ingredients to improve cognitive function, mood, well-being, and overall levels of affects are largely undetermined. The purpose of this study is to determine the effects of a combination of two dietary supplements, Scutellaria baicalensis and Acacia catech, on cognitive function, well-being, mood, cognitive interferences, and inflammation.

DETAILED DESCRIPTION:
The proposed study design will be a randomized, double-blind, placebo-controlled, parallel design to evaluate the effect of the supplement on cognitive function, well-being, mood, cognitive interferences, and inflammation. Participants will complete a series of psychological questionnaires, cognitive assessments, and venous blood draws.

Screening Visit (Visit 1) Upon arrival to the lab, participants will receive an informed consent document and will be required to give full consent before proceeding. Upon providing consent, participants will provide personal and emergency contact information before completing a health history form, exercise history form, and a physical activity questionnaire. Prior to this visit and each subsequent visit, participants will be required to observe an overnight fast (8-10 hours) of food or drink with calories including any foods or beverages that contain alcohol, caffeine, and nicotine. Participants will be instructed to be well-rested and to avoid exercise for 24 hours prior to each visit. Water intake will be encouraged during this time for appropriate hydration status. Participants will then have their height, body mass, resting heart rate, blood pressure, and urine specific gravity measured prior to completing their body composition assessment (only study visit 1) using a bioelectrical impedance analyzer (BIA). This study visit and all subsequent study visits will be scheduled between 0600 - 1000 hours. This study visit is estimated to take about 45 minutes to complete.

Visit 2-4 There is no required minimum time between Visit 1 and Visit 2. Visit 3 will occur 15 ± 3 days after Visit 2, 2 and Visit 4 will occur 28 ± 3 days after Visit 3. Participants will be required to follow identical pre-testing guidelines consisting of an overnight fast (8-10 hours) of food or drink with calories including any foods or beverages that contain alcohol, caffeine, and nicotine. Participants will be instructed to be well-rested and to avoid exercise for 24 hours prior to each visit. Water intake will be encouraged during this time for appropriate hydration status. Body mass, resting heart rate, and resting blood pressure will be measured. Female participants will take a urine pregnancy test to ensure they are not pregnant. Using standard phlebotomy approaches, approximately 21 mL of venous blood will be collected from a forearm vein. Participants will then complete the NIH Toolbox Cognitive Function Battery, NIH Toolbox Emotion Function Test, RAND SF-36 to assess well-being/mood, Stroop Color and Word test, Trail Making Test A and B, Finger tapping test, and the NIH Toolbox General Life Satisfaction score. After baseline testing, participants will be randomly assigned in a double-blind fashion to ingest on a daily basis for 6 weeks either a placebo or a dietary supplement. They will consume their supplement at the end of visits 2 and 3. Supplement compliance will be assessed through daily logging by the participant and checked by research team members calculating remaining amount of supplement during study visits.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult participants who are 30 to 60 years of age (inclusive).
2. In good general health (no active or uncontrolled diseases or conditions).
3. Have a body mass index (BMI) between 18.0 to 34.9 kg/m2 (inclusive).
4. Have normal or acceptable to the investigator vital signs (blood pressure and heart rate) at screening and/or baseline.
5. Individuals with childbearing potential must agree to practice an acceptable form of birth control for a certain timeframe prior to the first dose of study product and throughout the study, including:

   1. use for at least 3 months prior to the first dose of study product: hormonal contraceptives including oral contraceptives, hormone birth control patch (e.g., Ortho Evra), vaginal contraceptive ring (e.g., NuvaRing), injectable contraceptives (e.g., Depo-Provera, Lunelle), or hormone implant (e.g., Norplant System); or
   2. use for at least 1 month prior to the first dose of study product: double-barrier method, intrauterine devices, or complete abstinence from sexual intercourse that can result in pregnancy; or
   3. vasectomy of partner at least 6 months prior to the first dose of study product.

   Individuals with the potential to impregnate others must agree to use condoms or other acceptable methods to prevent pregnancy throughout the study. Complete abstinence from sexual intercourse that can result in pregnancy is also acceptable.
6. Agree to refrain from treatments listed in Section 6.4 in the defined timeframe.
7. Willing to refrain from changing their diet or lifestyle significantly for the duration of the study.
8. Willing and able to agree to the requirements and restrictions of this study, be willing to give voluntary consent, be able to understand and read the questionnaires, and carry out all study-related procedures.

Exclusion Criteria:

* 1. Participants who are lactating, pregnant or planning to become pregnant during the study.

  2. Have a known sensitivity, intolerability, or allergy to any of the study products or their excipients, or any of the rescue medications.

  3. Received a vaccine for COVID-19 in the 2 weeks prior to screening or during the study period, current COVID-19 infections, or currently have the post COVID-19 condition as defined by World Health Organization (WHO) (i.e., individuals with a history of probable or confirmed SARS-CoV-2 infection, usually 3 months from the onset of COVID-19 with symptoms that last for at least 2 months and cannot be explained by an alternative diagnosis).

  4. Participants with diagnosed type I or type II diabetes. 5. Having a history of heart disease, uncontrolled high blood pressure (≥140 mmHg systolic or ≥90 mmHg diastolic), renal or hepatic impairment/disease, major affective disorders, hepatic or renal dysfunction, unstable thyroid disease, immune disorders and/or immunocompromised (e.g. HIV/AIDS), cognitive impairment, neurological condition, or neurological disease, psychiatric disorder that required hospitalization in the past year, cancer (except localized skin cancer without metastases or in situ cervical cancer) within 5 years prior to the screening visit, or any clinically significant disease or disorder which, in the opinion of the investigator, may either put the potential participant at risk because of participation in the study, or influences the results or the potential participant's ability to participate in the study.

  6. Major surgery in 3 months prior to screening or planned major surgery during the course of the study.

  7. Participant has a pacemaker or implantable cardiac defibrillator. 8. Participant has an abnormality or obstruction of the gastrointestinal tract precluding swallowing (e.g. dysphagia) and digestions (e.g. known intestinal malabsorption, celiac disease, inflammatory bowel disease, chronic pancreatitis, steatorrhea).

  9. Participant has a history of alcohol or substance abuse in the 12 months prior to screening.

  10. Receipt or use of test product(s) in another research study within 28 days prior to baseline or longer if the previous test product is deemed by the investigator to have lasting effects that might influence the eligibility criteria or outcomes of current study.

  11. Any other active or unstable medical conditions or use of medications/supplements/ therapies that, in the opinion of the investigator, may adversely affect the participant's ability to complete the study or its measures or pose a significant risk to the participant.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2022-06-03 (Actual); Primary Completion 2022-10-18 (Actual); Study Completion 2022-10-18 (Actual)

PRIMARY OUTCOMES:
NIH Toolbox Cognitive Testing - Flanker Inhibitory Control | 30 days
  The first test is the Flanker inhibitory control and attention test which tests the participant's attention and executive function. This test requires the participant to maintain attention on a central stimulus while inhibiting the attention to distracting stimuli. The participant will be asked to match the direction of the central arrow while disregarding the surrounding distraction arrows. This test will measure both the reaction time and the accuracy of the participant's decisions.
NIH Toolbox Cognitive Testing - dimensional change card sort test | 30 days
  The second test is the dimensional change card sort test which measures a component of executive function known as set-shifting. Set-shifting is the ability to change responses based on a set of rules. In this test the participant will match images based either on color or shape. This test will measure both the reaction time and the accuracy of the participant's decisions.
  The third test is the pattern comparison processing speed test which measures processing speed. The participants will be shown two images and will be asked to evaluate if they are the same image. This test will measure the number of items that are answered correctly in 85 seconds.
NIH Toolbox Cognitive Testing - Pattern Comparison Processing Speed Test | 30 days
  The third test is the pattern comparison processing speed test which measures processing speed. The participants will be shown two images and will be asked to evaluate if they are the same image. This test will measure the number of items that are answered correctly in 85 seconds.
NIH Toolbox General Life Satisfaction Questionnaire | 30 days
  The NIH Toolbox was created to standardize the measure of positive and negative aspects of emotions.6 The effect of the study product on the participants' life will be measured using the general life satisfaction questionnaire from the NIH Toolbox. This will measure the participant's satisfaction with themselves and other areas of their life.6 This questionnaire will be completed on Visits 2, 3, and 4.
RAND SF-36 Questionnaire | 30 days
  The RAND SF-36 is a short questionnaire that measures health-related quality of life.7 The questionnaire measures eight concepts of health using 36 questions.7 The eight concepts measured are: physical functioning, pain, role limitations due to physical health, role limitations due to emotional problems, emotional well-being, social functioning, energy/fatigue, and general health. This questionnaire will be completed on Visits 2, 3, and 4.
Stroop Color Test | 30 days
  The Stroop color test measures the ability to stop cognitive interference of processing an initial stimulus from interfering with the simultaneous processing of a second stimulus.8 The participant will be tested using an app (Brain Test - Stroop Effect, Attila Hegedus, v1.5.0) on a tablet (iPad, Apple, Inc.). In a seated positions with no other distractions, the participant will be shown two color words, red or green. The words could be written in congruent conditions (e.g., the word red written in red ink) or incongruent conditions (e.g., the word red written in green ink). The participant must select the correct matching ink color for the presented word. The participant will have 60 seconds to match as many conditions correctly as possible. Correct responses add one point and incorrect responses will subtract one point from the total score. The test will be repeated three times and the best score will be recorded. This test will be completed on Visits 2, 3, and 4.
Trail Making Test Parts A & B | 30 days
  The trail making test provides information of cognitive processes such as attention, flexibility, and visual search and scanning.9 The participant will be tested using an app (INPL Trail Making Test, Motus Design Group) on a tablet (iPad, Apple, Inc.) in a comfortable seated position. When conducting the test there are two parts, part A and B. Part A requires the participant to tap circled numbers in sequence as quickly as possible (i.e., 1-2-3, etc.). Part B requires the participant to tap both circled numbers and letters in alternating numeric and alphabetical order as quickly as possible (i.e., 1-A-2-B, etc.). The time that it takes to complete each part of the test will be measured. This test will be completed on Visits 2, 3, and 4.
Finger Tapping Test | 30 days
  The finger tapping test is commonly used to evaluate the motor function and muscle control of the upper extremities.10 The participant will be tested using an app (Finger Tapping Test, SYBU Data, v3.5) on a tablet (iPad, Apple, Inc.). They will be instructed to sit comfortably in a chair with their palm flat on a desk or table. In this position, the participant will begin the test by tapping on the screen with the index finger of their dominant hand as quickly and consistently as they can in 10 second intervals. The participant will get one practice trial before completing three consecutive trials. Approximately 30 seconds of rest will be given in between each practice and testing trial. After the dominant hand is tested, the participant will repeat the test using the non-dominant hand. Upon completion of the third trial, the average number of taps for both the dominant and non-dominant hand will be calculated and recorded. This test will be completed on Visits 2, 3, and 4

SECONDARY OUTCOMES:
Blood Collection - C-Reactive Protein (CRP) | 30 days
  CRP is a non-specific indicator for inflammation. Studies have shown that there is an association between elevated levels of CRP and an increased risk of dementia and cerebrovascular disease in clinically compromised populations.
Blood Collection - Cortisol | 30 days
  Both dementia and mild cognitive impairment have been associated with elevated levels of cortisol. Chronic elevated levels of cortisol cause functional atrophy to areas of the brain that are associated with cognitive function.
Blood Collection - Brain Derived Neurotrophic Factor (BDNF) | 30 days
  BDNF is essential in the function of neural processes, and changing levels may contribute neurodegenerative diseases. In conditions of low BDNF there is growing evidence to show that the brain is more susceptible to oxidative stress.
Blood Collection - Uric Acid | 30 days
  Uric acid is a natural antioxidant and contributes greatly to the antioxidant capabilities of blood plasma. Increased oxidative stress has been associated with increased risk of cognitive impairment and dementia.
Resting Heart Rate | 30 days
  5 minute resting heart rate taken
Resting Blood Pressure | 30 days
  5 minute resting blood pressure taken

CONTACTS AND LOCATIONS:
Locations (1):
- Exercise and Performance Nutrition Laboratory, Saint Charles, Missouri, United States

IPD SHARING:
Plan to Share IPD: No